CLINICAL TRIAL: NCT06273137
Title: Mitigating Depression Among Adversity Exposed Adolescents Using Positive Affect Therapy
Brief Title: Positive Affect Treatment for Adolescents with Early Life Adversity
Acronym: PAT4ELA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Kate Kuhlman, Associate Professor, University of California, Irvine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2963
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either receive PAT or one of two control conditions (waitlist, supportive psychotherapy) upon enrollment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Positive affect treatment (Experimental): PAT is a 15-week cognitive-behavioral therapy that focuses on increasing reward motivation and sensitivity at the neural, behavioral, and affective levels of analysis. These observed effects occur through PAT's effects on reward sensitivity and positive affect. Participants will be assigned to a therapist with training in cognitive-behavioral therapy who will meet with them weekly via telehealth.
  Interventions: Behavioral: Positive affect treatment
- Waitlist (No Intervention)
- Supportive Psychotherapy (SUP) (Active Comparator): Participants randomized to SUP will receive 15 weeks of SUP from a doctoral student in clinical psychology. SUP is a flexibly-delivered, manualized evidence-based treatment that focuses on reinforcing a patient's existing coping strategies while fostering a positive therapeutic relationship. Supportive psychotherapy provides a time, attention, and social support control that is similar to a placebo but likely to be perceived as relevant to this population.
  Interventions: Behavioral: Supportive psychotherapy (SUP)

INTERVENTIONS:
Behavioral: Positive affect treatment — PAT includes 15 weekly, 1-hour sessions. The treatment is composed of three modules targeting behaviors (Sessions 1-7), cognitions (Sessions 8 -10), and compassion (Sessions 11-14), with skills being reinforced in a cumulative manner in subsequent sessions. The final session in the original treatment (Session 15) addressed relapse prevention, which will be adapted to focus on further reinforcing and generalizing learned skills. The treatment includes guided activities that target different aspects of positive affectivity such as reward approach-motivation, reward learning, and reward attainment.
  Other Names: PAT
  Arms: Positive affect treatment
Behavioral: Supportive psychotherapy (SUP) — Supportive psychotherapy provides a time, attention, and social support control that is similar to a placebo but likely to be perceived as relevant to this population.
  Arms: Supportive Psychotherapy (SUP)

SUMMARY:
Youth exposed to early life adversity (ELA) are known to be at greater risk for depression and suicidality and account for almost half of the youth suffering from psychiatric diseases today. Youth exposed to ELA consistently report symptoms of anhedonia as well as dysregulated positive affect. The present project will test the efficacy of PAT in a sample of ELA-exposed adolescents in order to determine whether PAT increases positive affect, and subsequently symptoms of depression. For the initial pilot phase of the investigation, the investigators will recruit up to 30 adolescents exposed to two or more childhood adversities (ACEs) who do not currently have major depressive disorder, and randomize them (1:1) to either participate in PAT or a waitlist control condition. For the second phase of the investigation, the investigators will recruit up to 300 adolescents exposed to two or more childhood adversities (ACEs) who do not currently have major depressive disorder, and randomize them (1:1) to either participate in PAT or supportive psychotherapy. For both phases, at study enrollment, then 4-, 8, and 12-months thereafter the investigators will measure positive affect and depressive symptoms (including anhedonia and reward sensitivity). The results of this study will be used to inform whether PAT has the potential to prevent major depressive episodes among adversity-exposed youth.

ELIGIBILITY:
Inclusion Criteria:

* aged 12-16
* exposed to 2 or more adverse childhood experiences (ACEs)

Exclusion Criteria:

* currently taking an antidepressant or any medications known to influence immune functioning on a daily basis (e.g., steroidal medications to treat asthma or allergies)
* current or past history of manic or psychotic symptoms
* parent-reported diagnosis of intellectual disability or autism spectrum disorder
* chronic medical conditions (e.g., cancer, rheumatoid arthritis, diabetes, multiple sclerosis),
* bleeding disorders such as hemophilia

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2024-02-03 (Actual); Primary Completion 2030-10-31 (Estimated); Study Completion 2030-10-31 (Estimated)

PRIMARY OUTCOMES:
depressive symptoms - anhedonia subscale | 4 months / end of treatment
  Reynolds Adolescent Depression Scale 2nd Edition - anhedonia subscale score; Scores can range from 7-28 with higher values indicating more severe anhedonia.
reward sensitivity | 4 months / end of treatment
  Reward motivation will be assessed behaviorally with the Effort Expenditures for Reward Task (EEfRT). The EEfRT assesses reward sensitivity by compelling participants to choose to engage in high and low effort motor tasks for varying potential monetary gains and computes reward sensitivity as the difference in propensity to choose hard choice trials at increasing trial values.
Systemic inflammation - C-reactive protein (CRP) | 4 months / end of treatment
  C-reactive protein concentrations measured in saliva; assay detection range is approximately 25 pg/mL - 1600 pg/mL with higher values indicating the presence of more systemic inflammation.

SECONDARY OUTCOMES:
Inflammatory gene expression | 4 months / end of treatment
  Degree of expression of 19 pro-inflammatory genes as measured via genome-wide transcriptional profiling of RNA from peripheral blood mononuclear cells. Values are expressed as z-scores, and higher values indicate greater average expression of pro-inflammatory genes.

OTHER OUTCOMES:
Positive affect | 4-months / end of treatment
  Positive and negative affect Schedule (PANAS) - positive affect subscale score; scores can range from 10 to 50 with higher values indicating more positive affect.
depressive symptoms - total | 4 months / end of treatment
  Reynolds Adolescent Depression Scale 2nd Edition (RADS-2) - Total Score; Scores can range from 30-120 with higher values indicating more depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Kate R Kuhlman, Principal Investigator — UC Irvine
Locations (1):
- University of California Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared with other researchers.